CLINICAL TRIAL: NCT01366560
Title: A Double Blind Randomised Placebo Controlled Two Way Cross Over Study to Determine the Effect of GSK962040 on Oesophageal Function and Gastric Emptying in Healthy Male Volunteers.
Brief Title: Effect of GSK962040 on Oesophageal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114639
Record Dates: First submitted 2011-02-03; First posted 2011-06-06 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Gastrointestinal Motility
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK962040 (Experimental): The subjects will be administered GSK962040 125 mg tablet as a single dose on Day 1 of study treatment visit. After 2 hours, the subjects will be administered wireless motility capsule. The subjects will be observed for expulsion of WMC in stool. Each subject will attend the clinical unit for two study treatment visits which will be separated by at least one week.
  Interventions: Drug: Active
- Placebo (Placebo Comparator): The subjects will be administered placebo tablet as a single dose on Day 1 of study treatment visit. After 2 hours, the subjects will be administered wireless motility capsule. The subjects will be observed for expulsion of WMC in stool. Each subject will attend the clinical unit for two study treatment visits which will be separated by at least one week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active — GSK962040 125mg
  Arms: GSK962040
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
GSK962040 is a selective non-peptide motilin receptor agonist which is in development for the treatment of conditions associated with slow rates of gastric emptying. Single ascending doses (1 to 150 mg), and 14-days repeated doses (10 to 125 mg daily) have been investigated in two randomized, placebo-controlled trials. Results show that these doses were well tolerated with few mild to moderate adverse events (AE), and no clinically significant abnormal vital sign measurements, ECG changes or abnormal clinical laboratory findings. GSK962040 exhibited predictable PK with and without food. The mean within subject time for half a [13C]-containing meal to empty from the stomach (GE t½) decreased by 22-43% from placebo with GSK962040 50-150 mg single doses, and shortening of gastric emptying was confirmed at doses of 50 mg and above in the repeat dose study.

Several studies have shown that motilin agonists increase lower oesophageal sphincter (LOS) pressure and have various dose dependent effects on oesophageal peristaltic amplitudes and propulsive contractions in both healthy volunteers and patients with gastro-oesophageal reflux disease (GORD). The purpose of the present study is to examine the effect of GSK962040 on oesophageal function, using techniques such as high resolution oesophageal manometry, and pH/gastric transit using a wireless motility capsule.

DETAILED DESCRIPTION:
Motilin is a peptide found in specific endocrine cells in the epithelia of the upper small intestine . It is released during fasting to act at its own receptor (motilin receptor, previously known as GPR38) resulting in the initiation of Phase III of the migrating motor complex (MMC). MMCs begin in the upper regions of the gut and are usually characterized by three distinct phases (I, a period of near-quiescence; II, short- or non-propulsive contractions at irregular frequency; III, a final burst of high amplitude propulsive contractions), terminating within the distal regions of the small intestine. Phase III activity may help clear the stomach and intestine from any undigested material, prevent bacterial overgrowth in the upper gut and perhaps help develop the sensation of hunger. The association of motilin release with Phase III of the MMC, together with an ability of motilin to mimic the strong propulsive contractions which comprise Phase III, has argued for an involvement of motilin in the regulation of certain functions of the gut during fasting.

Motilin receptor agonists can increase gastric emptying after ingestion of a meal; this action is mediated via the cholinergic system of the stomach. Erythromycin and motilides (non-peptide derivatives of macrolide antibiotics but devoid of antibiotic activity) are motilin receptor agonists and effective gastroprokinetic agents in patients. Erythromycin has been shown to stimulate gastric emptying in patients with diabetic, idiopathic and post-vagotomy gastroparesis, and in critically-ill patients receiving enteral nutrition, EM574 and KC 11458, and the peptide motilin receptor agonist atilmotin, also increase gastric emptying in humans.

In addition to effects on gastric emptying, motilin also appears to produce an effect on the oesophageal musculature. In particular, several studies have shown that single doses of motilin agonists (erythromycin in healthy volunteers and in patients with gastro-oesophageal reflux disease (GORD), atilmotin, a peptide motilin agonist, in healthy volunteers) , increase lower oesophageal sphincter (LOS) pressure and have various dose dependent effects on oesophageal peristaltic amplitudes and propulsive contractions in both healthy volunteers and patients with GORD. In addition, there is evidence that reduction of GORD in patients by using a motilin agonist may be useful clinically. For example, in a recent study in patients following lung transplantation, it was demonstrated that azithromycin, a motilin agonist macrolide antibiotic, reduced the number of reflux events and total oesophageal acid exposure as well as reduce the proximal extent to which reflux was regurgitated.

The clinical trials of promotility agents in GORD have not, however, shown consistent benefit. This may be related to compound characteristics. The dynamics of the relationship between PK and the effect on oesophageal function may be a factor as the most consistent data supporting their role as prokinetics in GORD come from studies which administered the drug intravenously, a route of administration which would not be suitable for a broader GORD population. In addition, if high doses of macrolides are required to have an effect on GORD, there is a risk of overlapping with antibiotic therapeutic doses, which would limit the interest of such approach. Macrolides also induce side effects such as nausea and abdominal, which makes macrolides difficult to tolerate for many patients. Another factor to consider is that repeat administration of macrolides induces desensitization of the motilin receptor reducing their efficacy over time, a phenomenon called tachyphylaxis. A strategy to decrease the tachyphylaxis to stimulation of motilin receptors is to identify agents that do not possess a complex motilide structure like erythromycin. This was the approach taken by GlaxoSmithKline (GSK) by which they identified GSK962040, a small molecule motilin receptor agonist, which is not a motilide.

GSK962040 was designed using the recombinant human motilin receptor to enhance the specificity for the receptor and potentially decrease the negative characteristics encountered with compounds with complex and non-specific motilide structures. A range of in vitro and in vivo studies have been conducted using GSK962040 to investigate its primary, secondary and safety pharmacology and toxicology. In addition, the pharmacokinetics (PK), absorption, distribution, metabolism and elimination of GSK962040 have been investigated in non-clinical species through a series of oral and intravenous studies.

The First Time in Human (FTIH) study (MOT107043) of GSK962040 is completed. It was an ascending single dose, randomised, placebo-controlled trial, with doses in the range of 1-150 mg to assess safety and tolerability, PK and pharmacodynamic effects on gastric emptying (GE) in healthy male and female volunteers. Dosing with GSK962040 was well tolerated. The results demonstrated that GSK962040 has an approximate dose proportional PK profile. Single doses of GSK962040 in the range of 1 to 150 mg resulted in mean exposures less than 23 μg.h/mL (AUC). At single doses of 50 mg to 150 mg, the rate of GE measured by the 13C-octanoic acid breath test was significantly increased in healthy volunteers when compared with placebo. Increasing the dose above 50 mg did not result in a greater effect on GE. The mean within subject time for half a [13C]-containing meal to empty from the stomach (GE t½) decreased by 22-43% from placebo with GSK962040 50, 75, 125 and 150 mg single doses (p ≤ 0.02). Increases in the rate of gastric emptying occurred in 85% to 100% of those healthy subjects receiving the 50 to 150 mg doses. The 14-day repeat dose study in healthy volunteers (MOT109681) was an ascending dose, randomised, placebo-controlled trial over the range of 10 mg to 125 mg daily. GSK962040 was well tolerated over the 14- day administration period for the doses tested and exhibited predictable PK, with and without food. The results indicated that GE was enhanced at doses of 50 mg and above, throughout the 14-day dosing. GSK962040 is currently in Phase II clinical development, being investigated in intensive care patients who receive enteral feeding, and in patients with diabetic gastroparesis. The present study will investigate effect of GSK962040 on oesophageal function because a combination of enhanced GE, barrier function (i.e. increase in LOS pressure) and oesophageal clearance would be potentially beneficial in patients with GORD or regurgitation.

Non clinical and clinical data indicate that a motilin agonist such as GSK962040 may also influence oesophageal function as well as GE. The purpose of the present study is primarily to evaluate the physiological effect of clinical doses of GSK962040 on oesophageal function in healthy volunteers, using established methods (oesophageal manometry, ambulatory pH/Impedance monitoring). GE will also be measured, using wireless motility capsule (WMC) monitoring. Given this is a physiological assessment, the use of healthy volunteers is considered appropriate; in addition, the study population will comprise male volunteers only in order to reduce variability in the measurements and therefore sample size, as GE varies with gender. The information from this study will inform decision making as to whether GSK962040 could have utility in conditions in which lower oesophageal function is deranged such as GORD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
3. AST, ALT, alkaline phosphatase and bilirubin = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
4. Subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication through at least 5 days following the dose of GSK962040.
5. Body weight = 50 kg and BMI within the range 18.5-29.9 kg/m2 (inclusive).
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. QTcB or QTcF < 450 msec or QTc<480msec in subjects with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
2. A positive test for HIV antibody.
3. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. History of cholecystectomy or biliary tract disease.
5. History of major gastrointestinal surgical procedure.
6. History of bowel surgery within the 3 months preceeding screening
7. History of strictures or adhesions following surgery.
8. History of, or current clinically significant gastrointestinal transit condition, ie. Passing of < 1 bowel movement per 48hr period.
9. A positive pre-study drug/alcohol screen.
10. A previous reaction or allergy to local anesthetic gels or sprays.
11. History of regular alcohol consumption within 6 months of the study defined as:

    -an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
12. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
13. Smoking history that includes regular use of tobacco or nicotine-containing products within 6 months prior to screening.
14. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
15. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
16. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
17. Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 90 day period.
18. Unwillingness or inability to follow the procedures outlined in the protocol.
19. Subject is mentally or legally incapacitated.
20. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2010-10-22 (Actual); Study Completion 2010-10-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline lower oesophageal sphincter (LOS) pressure (including pre and post prandial measures | Baseline and at 1hr30 and 2hr15mins post dose

SECONDARY OUTCOMES:
Change from baseline oesophageal peristaltic amplitudes | baseline and at 1hr30min and 2hr15mins post dose
Change from baseline oesophageal peristaltic velocity. | baseline and at 1hr30min and 2hr15mins post dose
Change from baseline proximal gastric pressure. | baseline and at 1hr30min and 2hr15mins post dose
Total gastric emptying time. | absolute transit time measured using SmartPill
Number and proximal extent of reflux episodes | 24hrs
Safety and tolerability of GSK962040 | baseline and at selected timepoints up to 24hrs post dose
  We will monitor ECG, vital signs, safety bloods and adverse events periodically throughout the study
Post prandial gastric and oesophageal pH | 2hr15mins post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hobson R, Farmer AD, Dewit OE, O'Donnell M, Hacquoil K, Robertson D, Barton ME, Dukes GE. The effects of camicinal, a novel motilin agonist, on gastro-esophageal function in healthy humans-a randomized placebo controlled trial. Neurogastroenterol Motil. 2015 Nov;27(11):1629-37. doi: 10.1111/nmo.12663. Epub 2015 Sep 8. PMID 26348542
- See also: Results for study 114639 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114639?search=study&search_terms=114639#rs
- Available data/document: Clinical Study Report: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114639 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register